CLINICAL TRIAL: NCT02785289
Title: A Comparison of Cotton and Flocked Swabs for Vaginal Self Collection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Manuela Viviano, Dr., University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2016-00412
Record Dates: First submitted 2016-05-17; First posted 2016-05-27 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Human Papillomavirus Infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flocked (Experimental): Patients will perform vaginal cell collection beginning with the flocked swab, followed by the coton swab.
  Interventions: Device: Vaginal swab
- Coton (Experimental): Patients will perform vaginal cell collection beginning with the coton swab, followed by the flocked swab.
  Interventions: Device: Vaginal swab

INTERVENTIONS:
Device: Vaginal swab — Vaginal cell collection will be performed with the two types of indicated swab.

SUMMARY:
The purpose of this study is to compare the performance of cotton and flocked swabs for vaginal self-sampling.

DETAILED DESCRIPTION:
Vaginal self-sampling for Human Papillomavirus (HPV) testing has been proposed as an efficient method cover hard-to reach populations in developing countries. While the recent cheap cotton swabs have traditionally been used for deoxyribonucleic acid (DNA) detection, recent studies have questioned their efficacy by reporting the superiority of the more expensive flocked swabs.

The objective of this study is to compare the performance of cotton vs flocked swabs for cellular retrieval and HPV DNA quantification after vaginal self-sampling.

A total of 120 women will be recruited. Inclusion criteria will be as follows: 21 years of age or older, attending the colposcopy clinic, understanding the study procedures and able to comply with the study protocol. Pregnant women, those having previously had a total hysterectomy, and women with ongoing menstruation will be excluded. Each woman will collect two different vaginal self samples: one with the cotton swab and one with the flocked swab. Subsequently, a flow cytometric analysis, as well as a real time PCR analysis and a cytologic evaluation for specimen adequacy will be run on each sample. Agreement between the two methods will be calculated using the kappa statistic (κ).

ELIGIBILITY:
Inclusion Criteria:

* attending the colposcopy clinic
* accepts voluntarily to take part to the study and signs the informed consent form

Exclusion Criteria:

* pregnancy
* previous hysterectomy
* ongoing menstruations

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Flow cytometric analysis | 1 week
  Number of epithelial cells
Real-time PCR analysis | 1 month
  HPV positivity

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided